CLINICAL TRIAL: NCT05500131
Title: The Association Between Restricted Ankle Joint Dorsiflexion and Dynamic Knee Valgus in Non-injured Youth Federated Basketball Players: a Cross-sectional Study
Brief Title: The Association Between Restricted Ankle Joint Dorsiflexion and Dynamic Knee Valgus
Acronym: TOBROD
Status: Completed | Type: Observational
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, CRISTINA ADILLÓN, Associate Professor, University Rovira i Virgili
Other Study IDs: 123/2018_3
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Knee Injuries; Ankle Injuries and Disorders; Movement, Abnormal; Adolescent Development
Keywords: Basketball; Adolescent; Knee valgus; Range of motion; Ankle
MeSH Terms: conditions — Knee Injuries; Ankle Injuries; Disease; Dyskinesias | interventions — Observation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: All participants allowed three practice trials for each test in this order: the Weight-bearing lunge test and the Single-leg squat test. Both of them were evaluated through the Leg Motion system (LegMotion, your MOtion®, Albacete, Spain)
  Interventions: Behavioral: Observation

INTERVENTIONS:
Behavioral: Observation — Ankle joint dorsiflexion was evaluated with the Weight-bearing lunge test through the Leg Motion system (LegMotion, your MOtion®, Albacete, Spain). Subjects were instructed to try to bring the knee to touch the metal rod (initially placed at a distance of 10 cm) without lifting the heel off the ground. The distance achieved was recorded in centimeters.
  Single-leg squat test was analyzed through the Leg Motion system (LegMotion, your MOtion®, Albacete, Spain). It consists of performing a monopodial squat to test dynamic knee valgus. They were to perform a single-leg squat to 30° knee flexion. The knee was considered to be aligned if the patella was over the second toe.

SUMMARY:
The purpose of this study was to analyze if a low ankle dorsiflexion range is associate with dynamic knee valgus in youth basketball players.

DETAILED DESCRIPTION:
Cross-sectional study. Ankle dorsiflexion range of motion was assessed by the Weight-bearing lunge test and the dynamic knee valgus by the Single leg squat test.

The participants were basketball players who belonged to youth basketball de-velopmental teams in the under-12 (U12), under-14 (U14), under-16 (U16) and under-17 (U17) categories. All participants were recruited by means of simple random sampling from the Catalan Basketball Federation during the 2018-2019 season. The participants were classified according to gender and age as stipulated by the rules determined an-nually for the respective official competitions. The study was carried out in the facilities of each club. The inclusion criteria were being age >12 and ≤17 at testing and actively competing during the study. Subjects were excluded if they had sustained any type of injury in the lower limbs before screening; presented any injury (overuse or acute) at the time of testing; if they had any oncological, psychological and/or psychiatric illnesses; or if they did not attend on the day of the assessment.

ELIGIBILITY:
Inclusion Criteria:

* Being age >12 and ≤17 at testing and actively competing during the study

Exclusion Criteria:

* Subjects were excluded if they had sustained any type of injury in the lower limbs before screening; presented any injury (overuse or acute) at the time of testing; if they had any oncological, psychological and/or psychiatric illnesses; or if they did not attend on the day of the assessment.

Ages: 12 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: The participants were basketball players who belonged to youth basketball de-velopmental teams in the under-12 (U12), under-14 (U14), under-16 (U16) and under-17 (U17) categories.
Sampling Method: Probability Sample
Enrollment: 791 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Ankle joint dorsiflexion | 1 year
  he Weight-bearing Lunge Test measured with the Leg Motion® system (Check Your Motion, Albacete) was used. Ankle dorsiflexion was recorded in centimeters.
Dynamic lower extremity valgus | 1 year
  The Single Leg Squat Test was used. The evaluator recorded a frontal and sagittal view with two filming devices. The knee was considered to be aligned if the patella was over the second toe.

SECONDARY OUTCOMES:
Age | 1 year
  Years
Age categories | 1 year
  According to the age of the participant could compete in 4 categories: U12, U14, U16 or U17.
Gender | 1 year
  Male or female
Weight | 1 year
  Kilograms
Height | 1 year
  Centimeters
Wingspan | 1 year
  Centimeters
Body mass index | 1 year
  Kg/m2
Hypermobility | 1 year
  Beighton's criteria (scores of >7 points out of a total of 9 points were considered hypermobile)

CONTACTS AND LOCATIONS:
Locations (1):
- Federación Catalana de Baloncesto, Barcelona, Spain